CLINICAL TRIAL: NCT06309719
Title: Characterizing the Healing of Periodontal Supra-bony Defects Treated With Hyaluronic Acid and Polynucleotides
Brief Title: Hyaluronic Acid and Polynucleotides for Supra-bony Defects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Geistlich Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 339479
Record Dates: First submitted 2024-02-16; First posted 2024-03-13 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Periodontal Diseases; Wound Heal; Periodontal Inflammation; Periodontal Pocket; Periodontal Attachment Loss
MeSH Terms: conditions — Periodontal Diseases; Periodontal Pocket; Periodontal Attachment Loss | interventions — Polydeoxyribonucleotides

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (Experimental): Periodontal Access Flap (AF) + Combined Formulation of Hyaluronic acid and Polydeoxyribonucleotides (PNHA)
  Interventions: Combination Product: Periodontal Access Flap (AF) + Combined Formulation of Hyaluronic acid and Polydeoxyribonucleotides (PNHA)
- Control (Active Comparator): Periodontal Access Flap (AF)
  Interventions: Procedure: Periodontal Access Flap (AF)

INTERVENTIONS:
Combination Product: Periodontal Access Flap (AF) + Combined Formulation of Hyaluronic acid and Polydeoxyribonucleotides (PNHA) — A conservative access flap will be performed such as simplified papilla preservation flap (SPPF). A PNHA gel will be placed on the root surfaces and supra-bony defects, followed by a tension-free primary closure of the interdental papillae and of the mucoperiosteal flaps by means of 5-0 suture
  Arms: Test
Procedure: Periodontal Access Flap (AF) — A conservative access flap will be performed such as simplified papilla preservation flap (SPPF). No gel will be placed before suturing the flap by tension-free primary closure of the interdental papillae and of the mucoperiosteal flaps by means of 5-0 suture
  Arms: Control

SUMMARY:
The goal of this pilot study is to describe the early wound healing molecular events and the vascularization pattern associated with the treatment of supra-bony defects with access flap alone or in association with a combined formulation of hyaluronic acid and polydeoxyribonucleotides gel.

DETAILED DESCRIPTION:
This is a parallel-group, pilot study aiming that consists of 7 visits over a minimum period of 4 months. Up to 24 periodontitis patients presenting with supra-bony defects will be recruited at the Centre for Oral Clinical Research (COCR) at the Institute of Dentistry, Barts and The London School of Medicine and Dentistry, Queen Mary University of London, United Kingdom.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy males and females ≥18 years old
* Stage III or IV periodontitis (Papapanou, Sanz et al. 2018)
* Presence of supra-bony periodontal defects (i.e., defects where the base of the pocket is located coronal to the alveolar crest and characterized by a predominantly horizontal pattern of tissue destruction) confirmed clinically and radiographically at a minimum of two and a maximum of four adjacent teeth and with a probing pocket depth (PPD) > 5 mm, following non-surgical periodontal therapy (NSPT). If >4 adjacent teeth exhibited the above clinical and radiographic conditions, the four adjacent teeth showing the greatest overall loss of periodontal attachment were included. Wisdom teeth and second molars will not be considered for the study.

If defect presents with an intrabony component, this should be ≤2 mm.

* Non-surgical periodontal treatment (step 1 and 2) completed within the previous 4 months
* Full-mouth bleeding score (FMBS) and full-mouth plaque score (FMPS) ≤20%

Exclusion Criteria:

* Teeth with degree III mobility
* Multi-rooted teeth with grade ≥2 furcation involvement
* Heavy smokers (≥10 cigarettes a day)
* Untreated caries or endodontic lesions or abscesses on the teeth involved in the surgery
* Previous periodontal surgery in the area selected for the study
* History of conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures (e.g., mitral valve prolapse, artificial heart)
* Antibiotic or anticoagulant therapy during the month preceding the baseline exam.
* History of alcohol or drug abuse
* Medical history that includes uncontrolled diabetes or hepatic or renal diseases, or other serious medical conditions that can have a negative impact on the periodontal condition
* In treatment with medications that can severely affect bone metabolism and blood clot formation (e.g., anticoagulants, long-term corticosteroids, bisphosphonates, immunosuppressants)
* Self-reported pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Early wound healing molecular events through GCF | Baseline, 1, 4, 7, 15 days and 3 months after surgery from the deepest site of one tooth involved in the surgery
  Characterize the early wound healing molecular events through gingival crevicular fluid (GCF) biomarkers. In particular, the expression of specific biomarkers involved in the recruitment of osteoblast precursors, inflammatory-immune response, organization of extracellular matrix, cell adhesion, oxidative stress and angiogenesis. Multiplex immunoassays will be employed to simultaneously assess the expression of multiple proteins in GCF samples on the biological processes involved in early periodontal wound healing and the mechanism of action of PNHA, focusing on the expression of specific signalling pathways, including but not limited to TNF alpha, NF-kappa B, IL-17, TGF-beta, VEGF, HIF-1, Chemokine and Wnt signalling pathways.
Early gingival tissue vascularization pattern when supra-bony defects are treated with AF, in association or not with PNHA | Before and straight after completing the surgery, as well as at day 1, 4, 7, 15 and at 3 months
  Blood flow changes in the surgical area will be evaluated with Laser Speckle Contrast Imaging (LSCI)

SECONDARY OUTCOMES:
Periodontal parameters and periodontal inflamed surface area (PISA) on the teeth involved in the surgery | Baseline and 3 months post-surgery
  PISA reflects the surface area of bleeding pocket epithelium in square millimetres. PISA is calculated using conventional clinical attachment levels (CAL), recession (REC) and bleeding on probing (BOP) measurements. PISA quantifies the amount of inflamed periodontal tissue, thereby quantifying the inflammatory burden posed by periodontitis. The higher the number, the more inflamed periodontal tissue. The periodontal inflamed surface area (PISA) is the sum of the PPD of bleeding on probing (BOP)-positive sites for the total dentition and can be easily calculated using routine periodontal charting.
Probing pocket depth (PPD) | Baseline and 3 months post-surgery
  PPD will be measured in mm using a University of North Carolina (UNC-15) periodontal probe at six sites per tooth/ implant (i.e., mesiobuccal, buccal, distobuccal, mesiolingual, lingual, and distolingual).
Gingival recession (REC) | Baseline and 3 months post-surgery
  REC will be measured in mm using a University of North Carolina (UNC-15) periodontal probe at six sites per tooth/ implant (i.e., mesiobuccal, buccal, distobuccal, mesiolingual, lingual, and distolingual).
Clinical attachment level (CAL) | Baseline and 3 months post-surgery
  CAL will be calculated considering the values for PPD and REC in mm
Suppuration | Baseline and 3 months post-surgery
  Suppuration will be recorded as percentage of total surfaces (6 aspects per tooth/implant), which reveal the presence of suppuration following periodontal probing. A binary score will be assigned to each surface (1 for suppuration present, 0 for suppuration absent).
Gingival phenotype | Baseline and 3 months post-surgery
  Gingival phenotype of the teeth involved in the surgery will be defined as thin (≤1.0 mm) or thick (>1mm) upon the observation of the periodontal probe through the gingival tissue
Keratinized tissue (KT) | Baseline and 3 months post-surgery
  Keratinized tissue width will be assessed in mm with a periodontal probe measuring from the mucogingival junction to the free gingival margin.
Full mouth plaque score (FMPS) | Baseline and 3 months post-surgery
  FMPS will be recorded as a percentage of total surfaces (6 sites per tooth/implant), which reveal the presence of plaque. A binary score will be assigned to each surface (1 for plaque present, 0 for absent).
Full mouth bleeding score (FMBS) | Baseline and 3 months post-surgery
  FMBS will be recorded as percentage of total surfaces (6 aspects per tooth/implant), which reveal the presence of bleeding within 10 - 30 seconds following periodontal probing. A binary score will be assigned to each surface (1 for bleeding present, 0 for bleeding absent).
Early Healing Index (EHI) | Day 1, 4, 7 and 15 after the surgical intervention
  The surgical wound will be graded as follows:
  1. complete flap closure - no fibrin line in the interproximal area
  2. complete flap closure - fine fibrin line in the interproximal area
  3. complete flap closure - fibrin clot in the interproximal area
  4. incomplete flap closure - partial necrosis of the interproximal tissue
  5. incomplete flap closure - complete necrosis of the interproximal tissue.
Gingival morphometric changes | Baseline visit, at 1, 4, 7, 15 days and 3 months post surgery
  An intra-oral 3D scanner will be used to capture and monitor soft tissue contour changes during early phase of healing. A series of subtracted images from the baseline to the subsequent follow-ups will accurately identify the area and magnitude of the swelling, changes in shape and volume to monitor/quantify the healing.
Oral impact on daily performance (OIDP) | Baseline and at 3 months post surgery
  OIDP focuses on the impact that the conditions of the teeth and mouth have on the physical (functional), psychological and social wellbeing of the person. For each performance, both the frequency and severity of oral impacts are assessed. The overall OIDP score ranges from 0 to 100, with higher scores indicating worse quality of life.
Dentine/root sensitivity | Baseline and at 3 months post-surgery
  A 100-mm horizontal visual analog scale (VAS) will be used to assess dentine/root sensitivity. The anchors for each end of the scales will be designated as none and extreme.
Food impaction | Baseline and at 3 months post-surgery
  A 100-mm horizontal visual analog scale (VAS) will be used to assess food impaction. The anchors for each end of the scales will be designated as none and extreme.
Patient perception about therapy | At day 1, 4, 7 and 15 after surgical therapy
  the extent of discomfort and/or pain experienced will be evaluated using a 100-mm VAS. The anchors for each end of the scales will be designated as none and extreme.
Global ratings of Periodontal Health and Quality of Life | 3 months after surgery
  Periodontal health and quality of life following periodontal therapy twill be investigated measured through specific questionnaries at 3 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Calciolari, DDS, MS, PhD, Principal Investigator — QMUL
Locations (2):
- United Kingdom (2):
  - Barts Health NHS Trust Dental Hospital, London
  - Centre for Oral Clinical Research (COCR), London